CLINICAL TRIAL: NCT04568993
Title: Patient-reported Outcome After Corticoid Injection for Triggerfinger- a Randomized Controlled Study Between Two Injection Procedures and Between Corticoid Injection and Percutaneous Release
Brief Title: The TriggerHappy Trial
Acronym: Triggerhappy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Joakim Stromberg, Senior consultant surgeon, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The TriggerHappy Trial
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Trigger Finger; Trigger Thumb; Minimally Invasive Surgery
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proximal phalangeal level (Experimental): injection in the the tendon sheet over proximal phalanx of finger
  Interventions: Procedure: Proximal phalangeal level
- volar MCP level (Active Comparator): injection above the A1 pulley volar to the MCP joint
  Interventions: Drug: Volar to the MCP-joint

INTERVENTIONS:
Procedure: Proximal phalangeal level — Injection of methyl prednisone and lidocaine in the tendon sheet at the level of the proximal phalanx
  Arms: proximal phalangeal level
Drug: Volar to the MCP-joint — Injection of methyl prednisone and lidocaine in the tendon sheet volar to the MCP-joint
  Arms: volar MCP level

SUMMARY:
This is a prospective randomized multicenterstudy focusing on PROMs after primary corticoid injection for triggerfinger with a comparison of two different injection techniques.

DETAILED DESCRIPTION:
This study aims to compare two different methods of corticosteroid injections in patients with triggerfinger, and to study the effects of these injections by day-to-day self-assessment by the included study persons for four weeks. The patient assess: 1. Pain 2. Motion and 3. Triggering by VAS scale every day for four weeks.

ELIGIBILITY:
Inclusion Criteria:•

1. Triggering of one or more fingers and/or impaired active finger motion and/or pain during active finger motion
2. Localized tenderness volar to the MCP joint of the affected finger
3. The patient seeks treatment

Exclusion Criteria:

1. Previous treatment for triggerfinger in the finger to be treated
2. Impaired function of finger due to previous trauma/infection or other condition
3. Suspicion of other cause than triggeriinger/tendovaginitis
4. Patient not able to follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain after injection | Four weeks
  Visual analouge scale (VAS), range 0-10, where 0 indicates "no pain" and 10 "maximum pain"
Impairment of finger motion | Four weeks
  Visual analouge scale (VAS), range 0-10, where 0 indicates "no impairment" and 10 "maximum impairment"
Triggering | Four weeks
  Visual analouge scale (VAS), range 0-10, where 0 indicates "no trigger phenomenon" and 10 "Trigger phenomenon all the time/ locked finger"

SECONDARY OUTCOMES:
Quick-DASH | Four weeks
  generic handquestionaire, 11 items, 0 means normal hand function, 100 most impaired function

CONTACTS AND LOCATIONS:
Locations (1):
- Alingsås Lasarett/ District Hospital, Alingsås, Sweden